CLINICAL TRIAL: NCT06333275
Title: Restoration of Immunity to Vaccine Preventable Diseases After CART-T Cell Therapy
Acronym: IMCAR
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: DLF-Nr: 5564; BASEC-Nr: 2023-01141 (Other: BASEC (Business Administration System for Ethics Committees) - Switzerland)
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Vaccine Immunity in CAR-T Cell Therapy Recipients
Keywords: CAR T-cell therapy; Vaccination
MeSH Terms: interventions — Tetanus Toxoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, EDTA-Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CAR T-cell recipients: Patients with B-cell malignancies receiving anti-CD19 or anti-BCMA CAR T-cell therapies
  Interventions: Biological: Vaccines against: Diphtheria, tetanus, pertussis, polio, haemophilus influenza type b, varicella and measles

INTERVENTIONS:
Biological: Vaccines against: Diphtheria, tetanus, pertussis, polio, haemophilus influenza type b, varicella and measles — First immunization course (6±1 months post CAR-T treatment):
  1. Diphtheria, tetanus, pertussis, polio, haemophilus influenza type b (as by the Swiss guidelines[FOPH] all of these are administered in one combined vaccine; INFANRIX DTPa-IPV+Hib Inj Susp®; GlaxoSmithKline)
  2. Hepatitis B (Engerix B®, GlaxoSmithKline)
  3. 13-valent Streptococcus pneumonia vaccine (Prevenar-13®; Pfizer)
  4. Herpes zoster vaccine in patients with documented prior seropositivity or known varicella-infection in patient history (as by The Swiss guidelines; Shingrix®; GlaxoSmithKline)
  5. Tick-borne encephalitis (as by The Swiss guidelines; FSME Immun CC®; Pfizer or Encepur N®, BavarianNordic; these vaccines can be used interchangeably)
  Second immunization course (12±1 months post CAR-T treatment):
  1. Mumps, measles, rubella (Priorix®, GlaxoSmithKline)
  2. Varicella zoster vaccine (as by guidelines; Varilrix®, GlaxoSmithKline) If seronegative/patient history negative

SUMMARY:
The goal of this observational study is to learn about vaccine immunity in patients with B-cell malignancies treated by chimeric antigen receptor T-cell therapies (CAR-T). The main questions it aims to answer are:

* Do CAR-T cell therapy recipients lose vaccine protection against common vaccine-preventable pathogens
* Are current re-vaccination recommendations sufficient in restoring vaccine-protection
* Is this restored vaccine-protection after CAR-T cell therapy lost faster than usual
* Do clinical or immunological factors predict vaccine response after CAR-T cell therapy

DETAILED DESCRIPTION:
B-cell malignancies are a diverse group of cancers that arise from abnormal growth and proliferation of B-cells, a type of cells that plays a crucial role in the immune system. The function of B-cells comprises the production of antibodies (immunoglobulins). Antibodies bind to specific molecules (antigens) on the surface of pathogens (e.g. viruses, bacteria) marking them for destruction by other components of the immune system. B-cell malignancies can arise from various stages of B-cell development and can manifest as a range of clinical presentations, from lymphomas with diverse clinical courses to aggressive leukemias. Treatment options for B-cell malignancies vary depending on the specific type of cancer and the stage of disease. Recently a broad array of newer immunotherapies became available[Feins 2019]. Specifically, the introduction of anti-CD19 and anti- BCMA (B cell maturation antigen) targeted chimeric antigen receptor T- cell therapy (CAR-T) represents a major treatment breakthrough in treatment of many B-cell malignancies[Sterner 2021, Haslauer 2021].

CAR-T therapy for B-cell malignancies involves extracting lymphocytes from a patient's blood and modifying them to produce chimeric antigen receptors (CARs) that can recognize and bind to proteins CD19 or BCMA expressed on cancer cells. The modified cells are then infused into the patient's bloodstream, where they seek out and bind to cancer cells expressing the target proteins. Once attached, the CAR-T cells are activated and initiate the destruction of the bound cancer cells. While CAR-T cell therapy has shown remarkable success in clinical trials[Sterner 2021, Haslauer 2021], it is a new and complex treatment with potential side effects such as cytokine release syndrome, neurotoxicity, and a significant impact on the host immune system[Kampouri 2022]. The tumor antigens targeted by CAR-T cells are also expressed on healthy B-cells (CD-19) and plasma-cells (BCMA). Therefore, CAR-T therapy leads to a decline in healthy B-cell populations with a subsequent decrease in antibody production (hypogammaglobulinemia)[Haslauer 2021]. The negative effects of CAR-T cell therapies on antibody concentrations leave individuals at risk of infection for a prolonged period[Wang 2020, Stewart 2021]. Currently, there is limited knowledge about the extent of loss of immunity against vaccine preventable diseases after CAR-T cell therapy[Kampouri 2022, Walti 2021]. High-quality evidence on how to prevent infections in CAR-T recipients and particularly on the necessity of re-vaccination against common vaccine-preventable pathogens, is lacking. Expert opinion statements recommend re-vaccinating these patients 6-12 months after CAR-T therapy against the most common pathogens[Hill 2020, Wudhikarn 2022]. Based on available recommendations and the vaccine-guidelines provided by the Swiss Federal Office of Public Health (FOPH) revaccination is started 6 months after CAR-T Therapy for inactivated vaccines and 12 months after CAR-T Therapy for life-attenuated vaccines.

With the present cohort study, the investigators aim to explore to which extent patients lose their humoral immunity to vaccine preventable pathogens after CAR-T cell therapies. Additionally, the investigators assess vaccine responses to routinely administered vaccinations in this population to examine whether re-vaccination after 6 months, as suggested in expert-opinion based recommendations[Hill 2020, Los-Arcos 2021] , is a reasonable approach. The vaccinations that are administered during the study period are usual care interventions according to published expert-opinion based guidelines[Hill 2020, Los-Arcos 2021, Plotkin 2010, FOPH]. These vaccines are presently administered to all CAR-T recipients at the University Hospital Bern and will be also administered to all CAR-T patients during the study period irrespective of study participation.

The results of this cohort study will reveal if present expert-opinion based vaccination recommendations for CAR-T patients are reasonable or if there will be need for adapting the recommendations (e.g. if it turns out that CAR-T patients do not lose protective immunity to vaccine preventable pathogens or if the study reveals that immunization according to present vaccine schedules do not elicit protective antibody levels). Furthermore, this project could increase fundamental understanding of immunological responses to common vaccines in the immunosuppressed population.

The present project falls into the risk category A according to art. 7 (HRO): It is a cohort study (no study intervention) with blood sampling (low risk sampling according to HRO art. 7.3.) Sampling includes minimal risk (e.g. hematoma after blood draw, uncomfortable feeling during procedure) for patients. Within this project, the investigators will exclusively use methods that are readily available in clinical practice (flow-cytometric analysis of lymphocyte populations, serology). Therefore, the gained knowledge will be immediately applicable in clinical practice and the results of this sub-project will help improving present vaccine strategies for CAR-T patients. Vaccination schedules are according to official recommendations by the Swiss Federal Office of Public Health and according to expert-opinion based guidelines and do not differ from patients not included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Suffering from a B-cell malignancy (B-cell acute lymphoblastic leukemia (ALL), B-cell non-hodgkin lymphoma (NHL), Follicular lymphoma (FL), Mantle Cell Lymphoma (MCL), Multiple myeloma (MM))
* Planned for a CAR-T cell therapy
* Provided written informed consent

Exclusion Criteria:

* Previous or already started CAR-T cell therapy
* < 18 years old
* Lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥ 18 years old) patients with B-cell malignancies (B-cell acute lymphoblastic leukemia, B-cell lymphoma, multiple myeloma) planned for CAR-T cell therapy at the oncology department of the University Hospital Bern, Switzerland will be prospectively included in the study.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
CAR-T cell therapy associated change in antibody levels against 5 vaccine preventable pathogens | 6 months after CAR-T cell therapy
  Change of antibody levels from baseline against tetanus, heamophilus type B, hepatitis B, poliovirus and measles virus after CAR-T cell therapy.

SECONDARY OUTCOMES:
Rate of seroprotection against tetanus 6 months after CAR-T cell therapy | 6 months after CAR-T cell therapy
  Rate of seroprotection against tetanus is assessed before re-vaccination. The investigators use cut-offs for protective antibody levels as previously defined by the FOPH and reported in the literature.
Rate of seroprotection against haemophilus influenza type B 6 months after CAR-T cell therapy | 6 months after CAR-T cell therapy
  Rate of seroprotection against haemophilus influenza type B is assessed before re-vaccination. The investigators use cut-offs for protective antibody levels as previously defined by the FOPH and reported in the literature.
Rate of seroprotection against hepatitis B virus 6 months after CAR-T cell therapy | 6 months after CAR-T cell therapy
  Rate of seroprotection against hepatitis B virus is assessed before re-vaccination. The investigators use cut-offs for protective antibody levels as previously defined by the FOPH and reported in the literature.
Rate of seroprotection against poliovirus 6 months after CAR-T cell therapy | 6 months after CAR-T cell therapy
  Rate of seroprotection against poliovirus is assessed before re-vaccination. The investigators use cut-offs for protective antibody levels as previously defined by the FOPH and reported in the literature.
Rate of seroprotection against measles virus 12 months after CAR-T cell therapy | 12 months after CAR-T cell therapy
  Rate of seroprotection against measles virus is assessed before re-vaccination. The investigators use cut-offs for protective antibody levels as previously defined by the FOPH and reported in the literature.
Rate of seroprotection against tetanus after re-vaccination following CAR-T cell therapy | 3-8 weeks after re-vaccination following CAR-T cell therapy
  Rate of seroprotection against tetanus after re-vaccination following CAR-T cell therapy. The investigators use cut-offs for protective antibody levels as previously defined by the FOPH and reported in the literature.
Rate of seroprotection against haemophilus influenza type B after re-vaccination following CAR-T cell therapy | 3-8 weeks after re-vaccination following CAR-T cell therapy
  Rate of seroprotection against haemophilus influenza type B after re-vaccination following CAR-T cell therapy. The investigators use cut-offs for protective antibody levels as previously defined by the FOPH and reported in the literature.
Rate of seroprotection against hepatitis B virus after re-vaccination following CAR-T cell therapy | 3-8 weeks after re-vaccination following CAR-T cell therapy
  Rate of seroprotection against hepatitis B virus after re-vaccination following CAR-T cell therapy. The investigators use cut-offs for protective antibody levels as previously defined by the FOPH and reported in the literature.
Rate of seroprotection against poliovirus after re-vaccination following CAR-T cell therapy | 3-8 weeks after re-vaccination following CAR-T cell therapy
  Rate of seroprotection against poliovirus after re-vaccination following CAR-T cell therapy. The investigators use cut-offs for protective antibody levels as previously defined by the FOPH and reported in the literature.
Rate of seroprotection against measles after re-vaccination following CAR-T cell therapy | 3-8 weeks after re-vaccination following CAR-T cell therapy
  Rate of seroprotection against measles virus after re-vaccination following CAR-T cell therapy. The investigators use cut-offs for protective antibody levels as previously defined by the FOPH and reported in the literature.
Clinical predictors of vaccine elicited immune response | Immediately before vaccination (6 months after CAR-T) and 4 weeks after vaccination (7 months after CAR-T)
  The investigators will explore whether certain patients factors (age, sex, type of cancer, previous autologous stem cell transplantation, previous anti-CD20 therapy) may be predictive for vaccine elicited immune responses 6 months post CAR-T treatment. The investigators will assess the correlation between mean fold-changes of vaccine elicited IgG concentrations (antibody concentration 4 weeks after vaccination: antibody concentration immediately before vaccination (6 months after CAR-T)) and the above mentioned predictor variables by regression analyses.
Immunological predictors of vaccine elicited immune response | Immediately before vaccination and 4 weeks after vaccination
  The investigators will explore whether certain immunological markers (counts of circulating CD19+ cells, CD4+ cells), and serum IgA concentration) measured immediately before vaccination at 6 months (for non-live vaccines) and 12 months (live vaccine) post CAR-T treatment may be predictive for vaccine elicited immune responses. The investigators will assess the correlation between mean fold-changes of vaccine elicited IgG concentrations (antibody concentration 4 weeks after vaccination(7 months after CAR-T): antibody concentration immediately before vaccination(6 months after CAR-T)) and the above mentioned immunological markers by regression analysis.
Persistence of vaccine elicited seroprotection | 13 months post CAR-T (7 months after vaccination with inactivated vaccines)
  The investigators will assess the proportion of patients with protective antibody titers at 13 months post CAR-T to each of following vaccine-preventable pathogens: tetanus, haemophilus influenza type B, hepatitis B, and poliovirus. The investigators use cut-offs for protective antibody levels as previously defined by the FOPH and reported in the literature.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Thurnheer Zürcher, PD, MD, Principal Investigator — University Hospital Bern, Switzerland; Cédric Hirzel, PD, MD, Principal Investigator — University Hospital Bern, Switzerland
Locations (1):
- University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Feins S, Kong W, Williams EF, Milone MC, Fraietta JA. An introduction to chimeric antigen receptor (CAR) T-cell immunotherapy for human cancer. Am J Hematol. 2019 May;94(S1):S3-S9. doi: 10.1002/ajh.25418. Epub 2019 Feb 18. PMID 30680780
- [Background] Sterner RC, Sterner RM. CAR-T cell therapy: current limitations and potential strategies. Blood Cancer J. 2021 Apr 6;11(4):69. doi: 10.1038/s41408-021-00459-7. PMID 33824268
- [Background] Haslauer T, Greil R, Zaborsky N, Geisberger R. CAR T-Cell Therapy in Hematological Malignancies. Int J Mol Sci. 2021 Aug 20;22(16):8996. doi: 10.3390/ijms22168996. PMID 34445701
- [Background] Wang Y, Liu Y, Tan X, Pan B, Ge J, Qi K, Cheng H, Cao J, Shi M, Yan Z, Qiao J, Jing G, Wang X, Sang W, Xia R, Zhang X, Li Z, Gale RP, Zheng J, Zhu F, Xu K. Safety and efficacy of chimeric antigen receptor (CAR)-T-cell therapy in persons with advanced B-cell cancers and hepatitis B virus-infection. Leukemia. 2020 Oct;34(10):2704-2707. doi: 10.1038/s41375-020-0936-4. Epub 2020 Jun 27. PMID 32594100
- [Background] Stewart AG, Henden AS. Infectious complications of CAR T-cell therapy: a clinical update. Ther Adv Infect Dis. 2021 Aug 24;8:20499361211036773. doi: 10.1177/20499361211036773. eCollection 2021 Jan-Dec. PMID 34457269
- [Background] Kampouri E, Walti CS, Gauthier J, Hill JA. Managing hypogammaglobulinemia in patients treated with CAR-T-cell therapy: key points for clinicians. Expert Rev Hematol. 2022 Apr;15(4):305-320. doi: 10.1080/17474086.2022.2063833. Epub 2022 Apr 11. PMID 35385358
- [Background] Walti CS, Krantz EM, Maalouf J, Boonyaratanakornkit J, Keane-Candib J, Joncas-Schronce L, Stevens-Ayers T, Dasgupta S, Taylor JJ, Hirayama AV, Bar M, Gardner RA, Cowan AJ, Green DJ, Boeckh MJ, Maloney DG, Turtle CJ, Hill JA. Antibodies against vaccine-preventable infections after CAR-T cell therapy for B cell malignancies. JCI Insight. 2021 Jun 8;6(11):e146743. doi: 10.1172/jci.insight.146743. PMID 33914708
- [Background] Hill JA, Seo SK. How I prevent infections in patients receiving CD19-targeted chimeric antigen receptor T cells for B-cell malignancies. Blood. 2020 Aug 20;136(8):925-935. doi: 10.1182/blood.2019004000. PMID 32582924
- [Background] Wudhikarn K, Perales MA. Infectious complications, immune reconstitution, and infection prophylaxis after CD19 chimeric antigen receptor T-cell therapy. Bone Marrow Transplant. 2022 Oct;57(10):1477-1488. doi: 10.1038/s41409-022-01756-w. Epub 2022 Jul 15. PMID 35840746
- [Background] Los-Arcos I, Iacoboni G, Aguilar-Guisado M, Alsina-Manrique L, Diaz de Heredia C, Fortuny-Guasch C, Garcia-Cadenas I, Garcia-Vidal C, Gonzalez-Vicent M, Hernani R, Kwon M, Machado M, Martinez-Gomez X, Maldonado VO, Pla CP, Pinana JL, Pomar V, Reguera-Ortega JL, Salavert M, Soler-Palacin P, Vazquez-Lopez L, Barba P, Ruiz-Camps I. Recommendations for screening, monitoring, prevention, and prophylaxis of infections in adult and pediatric patients receiving CAR T-cell therapy: a position paper. Infection. 2021 Apr;49(2):215-231. doi: 10.1007/s15010-020-01521-5. Epub 2020 Sep 26. PMID 32979154
- [Background] Plotkin SA. Correlates of protection induced by vaccination. Clin Vaccine Immunol. 2010 Jul;17(7):1055-65. doi: 10.1128/CVI.00131-10. Epub 2010 May 12. PMID 20463105
- See also: Swiss Federal Office of Public Health (FOPH) — https://www.bag.admin.ch/bag/de/home/das-bag/organisation/ausserparlamentarische-kommissionen/eidgenoessische-kommission-fuer-impffragen-ekif/impfempfehlungen.html